CLINICAL TRIAL: NCT01633476
Title: Does CMV Reactivation Cause Functional Impairment of CMV Specific CD4+ T-cells? The Potential for Valaciclovir to Prevent CMV-mediated Adverse Modulation of the Immune System in Patients With ANCA-associated Vasculitis
Brief Title: CMV Modulation of the Immune System in ANCA-associated Vasculitis
Acronym: CANVAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Professor Lorraine Harper (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor-Investigator, Professor Lorraine Harper, Professor of Nephrology, University of Birmingham
Organization: University of Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CMV-001; 097962/Z/11/Z (Other Grant/Funding Number: Wellcome Trust); 2012-001970-28 (EudraCT Number)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: ANCA Associated Vasculitis; CMV Infection
Keywords: CMV; ANCA associated vasculitis; CD4+CD28- T-cells; Valaciclovir
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Cytomegalovirus Infections | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valaciclovir (Active Comparator): Active treatment with valaciclovir
  Interventions: Drug: Valaciclovir
- No additional treatment (No Intervention): No additional treatment

INTERVENTIONS:
Drug: Valaciclovir — 2g q.d.s. orally for 6 months (dose adjusted according to renal function)
  Other Names: Brand names: Valtrex, Zelitrex
  Arms: Valaciclovir

SUMMARY:
The purpose of this study is to determine whether Cytomegalovirus (CMV) reactivation in ANCA-associated vasculitis (AAV) patients can be effectively and safely reduced using an antiviral agent (valaciclovir) and whether this in turn improves the function of the immune system thereby also improving the body's ability to fight other infections.

The primary hypothesis is that repeated episodes of CMV reactivation in AAV patients drive the expansion and functional impairment of CMV-specific T-cells, with increased susceptibility to infection. Inhibition of CMV replication with valaciclovir will block further stimulation of CMV specific T-cells and increase the functional capacity of the immune system.

DETAILED DESCRIPTION:
Infection is the commonest cause of death in patients with ANCA-associated vasculitis (AAV). The investigators have shown that the expansion of CD4+CD28- T-cells present in patients with AAV is driven by CMV and this expansion is associated with increased infection risk. It is suggested that these cells are driven by CMV reactivation and express markers of T-cell exhaustion with reduced cytokine production and inhibitory receptor expression. However the phenotype of CMV-specific T cells in those with extreme expansions of CD4+CD28- T-cells has not been explored.

The investigators aim to investigate the phenotype of CMV-specific T-cells comparing those patients with extreme expansions of CD4+CD28- T-cells to those with smaller expansions and relate this to CMV reactivation. The investigators will monitor CMV reactivation in urine and blood monthly by qPCR. This will be correlated with the expansion of CD4+CD28- T-cells and the phenotype of these cells, specifically looking at cytokine production and inhibitory receptor expression. The investigators will identify CMV-specific T-cells by MHC class II tetramers or by stimulating with CMV lysate. The investigators will proceed to undertake a randomised controlled trial with valaciclovir or no treatment to investigate whether the reduction of CMV reactivation improves the phenotype of CD4+CD28- T-cells in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Wegener's granulomatosis (now called Granulomatosis with Polyangiitis), microscopic polyangiitis or renal limited vasculitis according to Chapel Hill Consensus Conference criteria.
* In stable remission (no documented clinical disease activity) for at least 6 months prior to entry.
* On maintenance immunosuppression with prednisolone, mycophenolate mofetil or azathioprine alone or in combination (maximum 2 agents).
* Documented evidence of CMV infection (CMV-specific immunoglobulin G detected in peripheral blood).
* Documentation that female patients of child bearing potential are not pregnant and using an appropriate form of contraception.
* Written informed consent for study participation

Exclusion Criteria:

* Stage 5 chronic kidney disease (eGFR<15ml/minute/1.73m2).
* Other significant chronic infection (HIV, HBV, HCV, TB).
* B-cell or T-cell depleting therapy within 12 months.
* Treatment with anti-CMV therapies in last month
* Underlying medical conditions, which in the opinion of the Investigator place the patient at unacceptably high risk for participating in the study.
* Inability to fully or appropriately participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with CMV reactivation and time to CMV reactivation | Over 12 month period
  As assessed by measurable viral load on quantitative blood and urine CMV PCR.

SECONDARY OUTCOMES:
Proportion of patients experiencing adverse events sufficient to stop treatment | Over 6 month period (treatment period)
  Safety as defined by adverse events sufficient to stop treatment with trial drugs or serious adverse events and suspected unexpected serious adverse reactions (SUSARs).
Change in the proportion of the CD4+ CMV specific T cell population from baseline to 6 months | Baseline to 6 months
  Change in the proportion of CD3+CD4+CD28- T-cells
Change in markers of inflammation from baseline to 6 months | Baseline to 6 months
  Change in markers of inflammation including serum concentrations of pro and anti-inflammatory cytokines (TNF-a, IFN-g, IL-2, IL-6, IL-10, IL-17) and a marker of systemic inflammation (highly sensitive CRP).
Persistence of valaciclovir effect on proportion of CD4+ CMV-specific T cells at 6 months post treatment (i.e. change from 6 months to 12 months) | 6 months to 12 months
  Change in proportion of CD3+CD4+CD28- T-cells

OTHER OUTCOMES:
Change in the immune phenotype of the CD4+ and CD8+ T-cell compartment from baseline to 6 months | Baseline to 6 months
  Change in the proportion of naive and memory CD4+ and CD8+ T-cells
Change in the immune phenotype of CD4+ CMV-specific T-cells | Baseline to 6 months
  Change in cytokine production Change in inhibitory receptor expression

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Harper, MRCP PhD, Principal Investigator — University of Birmingham
Locations (1):
- Wellcome Trust Clinical Research Facility, Birmingham, United Kingdom

REFERENCES:
- [Background] Morgan MD, Pachnio A, Begum J, Roberts D, Rasmussen N, Neil DA, Bajema I, Savage CO, Moss PA, Harper L. CD4+CD28- T cell expansion in granulomatosis with polyangiitis (Wegener's) is driven by latent cytomegalovirus infection and is associated with an increased risk of infection and mortality. Arthritis Rheum. 2011 Jul;63(7):2127-37. doi: 10.1002/art.30366. PMID 21437878
- [Derived] Chanouzas D, Sagmeister M, Faustini S, Nightingale P, Richter A, Ferro CJ, Morgan MD, Moss P, Harper L. Subclinical Reactivation of Cytomegalovirus Drives CD4+CD28null T-Cell Expansion and Impaired Immune Response to Pneumococcal Vaccination in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. J Infect Dis. 2019 Jan 7;219(2):234-244. doi: 10.1093/infdis/jiy493. PMID 30102389
- [Derived] Chanouzas D, Dyall L, Nightingale P, Ferro C, Moss P, Morgan MD, Harper L. Valaciclovir to prevent Cytomegalovirus mediated adverse modulation of the immune system in ANCA-associated vasculitis (CANVAS): study protocol for a randomised controlled trial. Trials. 2016 Jul 22;17(1):338. doi: 10.1186/s13063-016-1482-2. PMID 27450392
- [Derived] Chanouzas D, Dyall L, Dale J, Moss P, Morgan M, Harper L. CD4+CD28- T-cell expansions in ANCA-associated vasculitis and association with arterial stiffness: baseline data from a randomised controlled trial. Lancet. 2015 Feb 26;385 Suppl 1:S30. doi: 10.1016/S0140-6736(15)60345-2. PMID 26312852